CLINICAL TRIAL: NCT04086563
Title: Effects of Motor Imagery in Pain Modulation and Median Nerve Mechanosensitive in Healthy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2703201906919
Record Dates: First submitted 2019-08-09; First posted 2019-09-11 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Median Nerve Injury
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Action observation (Experimental): The patients will observe a 25 minutes clip of neurodynamic exercises of the hand.
  Interventions: Other: Mirror therapy; Other: Neurodynamic exercises; Other: Strength
- Mirror Therapy (Experimental): With a mirror glasses, the patients will execute neurodynamic movements of their non-dominant hand during 25 minutes.
  Interventions: Other: Action observation; Other: Neurodynamic exercises; Other: Strength
- Strength Training (Active Comparator): Strength protocol for the dominant hand.
  Interventions: Other: Action observation; Other: Mirror therapy; Other: Neurodynamic exercises
- Neurodynamic exercise (Experimental): Active neurodynamic exercises for the dominant hand.
  Interventions: Other: Action observation; Other: Mirror therapy; Other: Strength

INTERVENTIONS:
Other: Action observation — look at a clip of a hand doing neurodynamic exercises.
  Arms: Mirror Therapy; Neurodynamic exercise; Strength Training
Other: Mirror therapy — With a mirror glasses on, do the neurodynamic exercises with the non-dominant hand while the patient is looking at the dominant hand
  Arms: Action observation; Neurodynamic exercise; Strength Training
Other: Neurodynamic exercises — active movement of the dominant hand. Do neurodynamic exercises.
  Arms: Action observation; Mirror Therapy; Strength Training
Other: Strength — Execute a short strength training for the dominant hand
  Arms: Action observation; Mirror Therapy; Neurodynamic exercise

SUMMARY:
The aim of this study are 1) to determinate the effectiveness of motor imagery or strength training in differens aspects of pain modulation. 2) evaluate the functional improvement of the hand by a motor imagery protocol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* be under 18
* any pathology which provoke pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-09-08 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Conditioned pain modulation | Change from baseline at 2 weeks
  Diffused noxious inhibitory control system will be measure with tourniquet test
Pressure pain threshold | Change from baseline at 2 weeks
  Three consecutive trials of pressure pain threshold on the active trigger point at a rate of 1 kg/sec at intervals of 30 seconds were conducted.
Cold hyperalgesia | Change from baseline at 2 weeks
  10 seconds of a cold pack and after that, rating the pain from 0 to 10
Neural mechanosensitive | Change from baseline at 2 weeks
  Upper Limb Neurodynamic test 1 (ULNT1)

SECONDARY OUTCOMES:
Strength_grip | Change from baseline at 2 weeks
  grip strength without pain
Imagine movement capacity | Change from baseline at 2 weeks
  testing the capacity of imagine that their own body is movement. Movement Imagery Questionnaire-Revised (MIQ-R questionaire).
  top score 56 and bottom score 8. The higher values indicates a better outcome.
Psychological factors_Anxiety | Change from baseline at 2 weeks
  State Trait Anxiety Inventory (STAI-T). Top score 60 and bottom score 0. The higher values indicate worst outcomes.
Psychological factors_Depression | Change from baseline at 2 weeks
  Beck Depression Inventory (BDI-II). the scores goes from 0 to 63. The higher values indicate worst outcomes.
  Beck Depression Inventory (BDI-II)
  Beck Depression Inventory (BDI-II)
Psychological factors_Kinesiophobia | Change from baseline at 2 weeks
  Tampa Scale for Kinesiophobia. Total scores goes from 11 to 44.The higher values indicate worst outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

REFERENCES:
- [Derived] Matesanz-Garcia L, Caceres-Pajuelo JE, Cuenca-Martinez F, La Touche R, Goicoechea-Garcia C, Fernandez-Carnero J. Effects of neural mobilizations through movement representation techniques for the improvement of neural mechanosensitivity of the median nerve region: a randomized controlled trial. Somatosens Mot Res. 2021 Dec;38(4):267-276. doi: 10.1080/08990220.2021.1964463. Epub 2021 Aug 17. PMID 34404324